CLINICAL TRIAL: NCT00168272
Title: A Randomised Double-Blind Trial of Low and High Frequency Stimulation rTMS (Repetitive Transcranial Magnetic Stimulation) In Major Depression
Brief Title: Priming rTMS In Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/04
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Last update posted 2007-04-16 (Estimated); Status verified 2007-04

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Magnetic Stimulation; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
The purpose of this study is to assist in understanding the most effective parameters for TMS in Depressive Disorders. Most research conducted has used high frequency stimulation on the left hemisphere.However, low frequency on the right hemisphere has also been shown to have antidepressant properties and appears to be better tolerated. A promising approach to improve responses to rTMS may be to combine high and low frequency stimulation where they are both applied to the right side of the brain. In this approach, high frequency stimulation is provided first which may 'prime' or pre-prepare the brain for low frequency stimulation in a way that enhances its response. Participants are randomised to receive active or placebo priming stimulation.If participants do not respond to this treatment condition after 10 sessions applied over a two week period they will be offered 10 session of high frequency left sided TMS treatment. Alternatively, if participants respond favorably they may continue with that treatment condition for another 10 sessions.

DETAILED DESCRIPTION:
The primary outcome measure used is the MADRS (Montgomery-Asberg Depression Rating Scale). This is administered at baseline and on a fortnightly basis. At study end response criteria is defined as a 50% reduction in total MADRS score and remission defined as a MADRS score of less than or equal to 10.

Other outcome measures administered fortnightly are: BPRS (Brief Psychiatric Rating Scale), CORE (measure of melancholic symptoms), BDI (Beck Depression Inventory), CGI (Clinical Global Impression Scale), GAF (Global Assessment of Functioning Scale). A cognitive battery is also administered.

Inclusion Criteria:

* Moderate to severe depressive symptoms as indicated as MADRS >20
* Failure to respond to a minimum of two antidepressant medications
* No increase or initiation of new antidepressant therapy in the four weeks prior to entering the trial Exclusion Criteria
* Have an unstable medical condition, neurological disorder or any history of seizure disorder or are currently pregnant or lactating
* Previous brain injury or surgery, any metal clips, plates or other metal items in the head, cardiac pacemaker
* In the opinion of the investigator, are a sufficient suicide risk to require immediate electro-convulsive therapy
* Have a current DSMIV diagnosis of substance abuse or dependence disorder, a diagnosis of a personality disorder or another axis 1 disorder

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe depressive symptoms as indicated as MADRS >20
* Failure to respond to a minimum of two antidepressant medications
* No increase or initiation of new antidepressant therapy in the four weeks prior to entering the trial

Exclusion Criteria:

* Have an unstable medical condition, neurological disorder or any history of seizure disorder or are currently pregnant or lactating
* Previous brain injury or surgery, any metal clips, plates or other metal items in the head, cardiac pacemaker
* In the opinion of the investigator, are a sufficient suicide risk to require immediate electro-convulsive therapy
* Have a current DSMIV diagnosis of substance abuse or dependence disorder, a diagnosis of a personality disorder or another axis 1 disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-06; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure used is the MADRS (Montgomery-Asberg Depression Rating Scale). At study end response criteria is defined as a 50% reduction in total MADRS score and remission defined as less or equal to 10.

SECONDARY OUTCOMES:
Other outcome measures administered fortnightly are: BPRS (Brief Psychiatric Rating Scale), CORE (measure of melancholic symptoms), BDI (Beck Depression Inventory), CGI (Clinical Global Impression Scale), GAF (Global Assessment of Functioning Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Fitzgerald, MBBS, PhD, Principal Investigator — Alfred Psychiatry Research Centre
Locations (1):
- Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia